CLINICAL TRIAL: NCT01562067
Title: Sonographic Characteristics of Tumor Indices in Patients With Cervical Cancer During Chemo-radiotherpy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 125-11CTIL
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2012-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Cancer
Keywords: Cervical tumors,vascular changes,Sonographic characteristics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — pap smear
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ultrasound examination — ultrasound and doppler studies to evaluate size and vascularity of tumor during radiotherapy
  Other Names: no other name

SUMMARY:
Cervical tumors are characterized by vascular changes (in terms of quantity, volume and Flows) in the tumor. Due to a good access to the cervix through the vagina, these parameters can be assessed using a three dimensional supersonic. Sonographic characteristics of tumor indices measures before and after oncological treatments may shed light on the patient's prognosis.

DETAILED DESCRIPTION:
no editional information. see above

ELIGIBILITY:
Inclusion Criteria:

* Cervical cancer patients intended to undergo chemotherapy or radiation, or both

Exclusion Criteria:

* no exclusions

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with cervical cancer during radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Sonographic characteristics of cervical tumors | 5 years
  Sonographic characteristics of cervical tumors indices measures before and after oncological treatments may shed light on the patient's prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: amnon amit, md, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel